CLINICAL TRIAL: NCT05114187
Title: An Internet-Based Education Program for Care Partners of People Living With Dementia (iGeriCare): A Pilot Randomized Controlled Trial
Brief Title: An Internet-Based Education Program for Care Partners of People Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: #21-24
Record Dates: First submitted 2021-10-15; First posted 2021-11-09 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Dementia; Burden, Caregiver; Self Efficacy; Knowledge
Keywords: Web-based intervention; Internet; E-health; Dementia; Caregiver; Alzheimer disease; Education and Training; Clinical Trial; Knowledge Translation
MeSH Terms: conditions — Dementia; Caregiver Burden; Alzheimer Disease | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: This study is a two-arm pilot randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Intervention (Experimental)
  Interventions: Other: Education Intervention
- Education Control (Active Comparator)
  Interventions: Other: Education Control

INTERVENTIONS:
Other: Education Intervention — Participants in the intervention group will be provided e-learning about dementia and promoting brain health, consisting of the following components:
  1. Ten selected multimedia e-learning lessons;
  2. A series of 16 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lessons.
  Participants will have 8-weeks to complete the intervention. The total time to complete is approximately 5-6 hours.
  Arms: Education Intervention
Other: Education Control — Participants in the control group will be provided e-learning about dementia and promoting brain health, consisting of the following components:
  1. One selected multimedia e-learning lesson;
  2. A series of 16 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lessons.
  Participants will have 8-weeks to complete. The total time to complete is approximately 1-2 hours.
  Note: All participants will receive access to all e-learning at the conclusion of the study.
  Arms: Education Control

SUMMARY:
With the aging population, the prevalence of dementia is increasing dramatically. People living with dementia are highly dependent on family care partners, who may have little knowledge of the disorder. National and provincial guidelines have all highlighted the importance of online resources to improve care partner education; however, very few have been widely implemented or rigorously studied.

The investigators have developed the award-winning dementia education platform to complement traditional patient and family educational approaches. It allows free access to multimedia e-learning lessons, live expert webinars, and email-based content that care partners can access any time, anywhere.

In a pilot randomized controlled trial (RCT), the investigators propose to study 1) the feasibility and care partner acceptance of the intervention and some of the study methods, and 2) the impact of the intervention on care partner self-efficacy, knowledge, and sense of burden.

This initiative has the potential to improve the quality, cost effectiveness, and efficiency of dementia care. The intervention could be easily scaled and spread both provincially and nationally to complement other dementia education methods, at a time when the prevalence of dementia is increasing and access to high quality internet-based interventions is essential.

ELIGIBILITY:
Inclusion Criteria:

1. they are a family and/or friend care partner of a person living with dementia,
2. they reside in Canada,
3. they are 18 years of age and over,
4. they have a good command of the English language,
5. they have access to email and internet,
6. they are comfortable using email and internet,
7. they have the ability to grant online informed consent, and
8. they complete online baseline assessments.

Exclusion Criteria:

1. they are a not family and/or friend care partner of a person living with dementia,
2. they do not reside in Canada,
3. they are not 18 years of age and over,
4. they do not have a good command of the English language,
5. they do not have access to email and internet,
6. they are not comfortable using email and internet,
7. they do not have the ability to grant online informed consent, and
8. they do not complete online baseline assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Intervention adherence (time spent) | 8 weeks
  Lesson completed data and email open rates will be collected and saved to quantify the time(s) spent on intervention activities.
Participant satisfaction | 8 weeks
  A custom satisfaction questionnaire data adapted from the Information Assessment Method For All (IAM4all) will be collected and saved to assess satisfaction with the intervention.
Participant satisfaction | 8 weeks
  A custom implementation oral interview questionnaire adapted from The Consolidated Framework for Implementation Research (CFIR) will be collected and saved to assess implementation of the intervention.

SECONDARY OUTCOMES:
Recruitment rates | 8 weeks
  Participant recruitment numbers will be collected and saved to quantify the number of interested participants.
Attrition rates | 8 weeks
  Participant attrition rates will be collected and saved to quantify the number of study dropouts vs completions
Change from baseline in the Revised Scale for Caregiving Self-Efficacy (RSCSE) at 8 weeks. | 0, 8 weeks
  Self-efficacy will be measured through the Revised Scale for Caregiving Self-Efficacy (RSCSE) (reliability α = >.80). The RSCSE contains 15 items within 3 subscales (self-efficacy for obtaining respite, responding to disruptive patient behaviours, and controlling upsetting thoughts about caregiving). Higher scores indicate a higher level of self-efficacy.
Change from baseline in the Dementia Knowledge Assessment Scale (DKAS) at 8 weeks. | 0, 8 weeks
  Knowledge will be measured through the Dementia Knowledge Assessment Scale (DKAS) (reliability α = .85; ωh = .87; overall scale). The DKAS consists of 25 items on different aspects of dementia that could be answered with 'True,' 'Probably True,' 'False, 'Probably False,' or 'I don't know.' Higher scores indicate a higher level of dementia knowledge.
Change from baseline in the Zarit Burden Interview (ZBI) at 8 weeks. | 0, 8 weeks
  Burden will be measured through the Zarit Burden Interview (ZBI) (reliability α = .92). The ZBI contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Higher scores indicate a higher level of burden.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Levinson AJ, Ayers S, Clark S, Woodburn R, Markle-Reid M, McKenna B, Oliver D, Papaioannou A, Siu H, Sztramko R. Web-Based Education Program for Care Partners of People Living With Dementia (iGeriCare): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 4;14:e67048. doi: 10.2196/67048. PMID 40466093